CLINICAL TRIAL: NCT00005757
Title: Racial Variation in ACE--Genetic and Physiologic Bases
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5115; R29HL056963 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover

SUMMARY:
To determine whether differences in the activity of the renin-angiotensin and bradykinin systems are involved in the pathogenesis of blood pressure variation in African Americans.

DETAILED DESCRIPTION:
BACKGROUND:

Each year, more than 40,000 new patients require treatment for end stage renal disease, a condition which is 4-fold higher among African Americans than Caucasians. Trials of angiotensin converting enzyme inhibitors (ACEIs) in Caucasians support a role of the renin-angiotensin system in the pathogenesis of glomerulosclerosis. Yet, despite the high prevalence of nephropathy among African Americans, Blacks have been under-represented in studies in ACEIs. Data from our laboratory suggest that the renal effects of ACEI may differ in African Americans. African Americans are resistant to the anti-hypertensive effects of ACEI and, thus, may be resistant to the renoprotective effects as well. The ACE deletion allele, a variant associated with increased ACE activity and progression of renal diseases, is increased in frequency in African Americans, while the frequency of the Ang AT1 receptor C allele, a variant associated with antihypertensive responsiveness to ACEI is decreased. Moreover, African Americans exhibit decreased sensitivity to Ang I and increased sensitivity to bradykinin. Taken together, these data suggest the hypothesis that ACE activity is increased in African Americans, leading to decreased bradykinin levels ( and receptor sensitization) and increased tissue Ang II (and receptor desensitization).

DESIGN NARRATIVE:

The study tests the hypothesis that ACE activity is increased in African Americans, leading to decreased bradykinin levels (and receptor sensitization) and increased tissue Ang II (and receptor desensitization). The effects of race, hypertension and ACE insertion/deletion genotype on ACE activity will be determined, as measured by the pressor and renal vasoconstrictor responses to Ang I and Ang II and the vasodilator response to bradykinin. Specific bradykinin and angiotensin receptor antagonists will be used to determine the relative contribution of increased bradykinin and decreased angiotensin II to the renal hemodynamic effects of ACEIs in African Americans and Caucasians.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 1997-09; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Brown — Vanderbilt University

REFERENCES:
- [Background] Brown NJ, Agirbasli MA, Williams GH, Litchfield WR, Vaughan DE. Effect of activation and inhibition of the renin-angiotensin system on plasma PAI-1. Hypertension. 1998 Dec;32(6):965-71. doi: 10.1161/01.hyp.32.6.965. PMID 9856958
- [Background] Gainer JV, Morrow JD, Loveland A, King DJ, Brown NJ. Effect of bradykinin-receptor blockade on the response to angiotensin-converting-enzyme inhibitor in normotensive and hypertensive subjects. N Engl J Med. 1998 Oct 29;339(18):1285-92. doi: 10.1056/NEJM199810293391804. PMID 9791144
- [Background] Murphey LJ, Hachey DL, Vaughan DE, Brown NJ, Morrow JD. Quantification of BK1-5, the stable bradykinin plasma metabolite in humans, by a highly accurate liquid-chromatographic tandem mass spectrometric assay. Anal Biochem. 2001 May 1;292(1):87-93. doi: 10.1006/abio.2001.5073. PMID 11319821
- [Background] Gainer JV, Brown NJ, Bachvarova M, Bastien L, Maltais I, Marceau F, Bachvarov DR. Altered frequency of a promoter polymorphism of the kinin B2 receptor gene in hypertensive African-Americans. Am J Hypertens. 2000 Dec;13(12):1268-73. doi: 10.1016/s0895-7061(00)01215-2. PMID 11130770
- [Background] Murphey LJ, Kumar S, Brown NJ. Endogenous bradykinin and the renin and pressor responses to furosemide in humans. J Pharmacol Exp Ther. 2000 Nov;295(2):644-8. PMID 11046100
- [Background] Brown NJ, Nakamura S, Ma L, Nakamura I, Donnert E, Freeman M, Vaughan DE, Fogo AB. Aldosterone modulates plasminogen activator inhibitor-1 and glomerulosclerosis in vivo. Kidney Int. 2000 Sep;58(3):1219-27. doi: 10.1046/j.1523-1755.2000.00277.x. PMID 10972684
- [Background] Murphey LJ, Gainer JV, Vaughan DE, Brown NJ. Angiotensin-converting enzyme insertion/deletion polymorphism modulates the human in vivo metabolism of bradykinin. Circulation. 2000 Aug 22;102(8):829-32. doi: 10.1161/01.cir.102.8.829. PMID 10952948
- [Background] Murphey LJ, Hachey DL, Oates JA, Morrow JD, Brown NJ. Metabolism of bradykinin In vivo in humans: identification of BK1-5 as a stable plasma peptide metabolite. J Pharmacol Exp Ther. 2000 Jul;294(1):263-9. PMID 10871321
- [Background] Wilsdorf T, Gainer JV, Murphey LJ, Vaughan DE, Brown NJ. Angiotensin-(1-7) does not affect vasodilator or TPA responses to bradykinin in human forearm. Hypertension. 2001 Apr;37(4):1136-40. doi: 10.1161/01.hyp.37.4.1136. PMID 11304515